CLINICAL TRIAL: NCT01469117
Title: Enteral Formula Tolerance In Pediatric Patients With Developmental Disabilities
Brief Title: Feeding Trial in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.03.US.HCN
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Developmental Disabilities
Keywords: Developmental disabilities; Enteral Nutrition; Tube feeding; Nutrition support
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric developmental disabilities: Children aged 1-13 years old with development disabilities, requiring enteral tube feeding for at least 14 days
  Interventions: Other: enteral formula

INTERVENTIONS:
Other: enteral formula — Complete feeding of study enteral formula, route and regimen prescribed by the physician

SUMMARY:
This is a single center, prospective, non-randomized, uncontrolled, observational study of the use of an enteral nutrition product in pediatric patients with developmental disabilities.

DETAILED DESCRIPTION:
This prospective observational study seeks to assess ability to achieve enteral feeding goals with a new tube feeding product in pediatric patients with developmental disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 1-13 years old with development disabilities
* Currently tolerating enteral feeding
* Requiring nutritional management to meet 50-90th% weight for age on the Kennedy Kreiger Growth Charts
* Requires enteral tube feeding for at least 14 days.

Exclusion Criteria:

* Unable to access gastrointestinal tract for feeding via tube
* Other condition which contraindicates tube feeding

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with developmental disabilities
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to feeding goal achievement | up to 14 days

SECONDARY OUTCOMES:
Gastrointestinal measures assessment | up to 21 days
Percentage of nutrition goal met | daily up to 21 days
Serum biochemical markers assessment | baseline and completion of study
Assessment of frequency and nature of adverse events | daily up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Darin Brannan, MD, Principal Investigator — The Children's Center
Locations (1):
- The Children's Center, Bethany, Oklahoma, United States